CLINICAL TRIAL: NCT00517803
Title: Micronutrient Supplemented Probiotic Yogurt for HIV/AIDS and Other Immunodeficiencies: A Randomized, Placebo-controlled Trial
Brief Title: Micronutrient Supplemented Probiotic Yogurt for HIV/AIDS and Other Immunodeficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-07-220; 13468
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections; Cancer, Second Primary
Keywords: micronutrients; immunodeficiency; probiotics; yogurt; Healthy; Acquired Immunodeficiency Syndrome; Complementary Therapies
MeSH Terms: conditions — HIV Infections; Neoplasms, Second Primary; Immunologic Deficiency Syndromes; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Probiotic Yogurt B: with various micronutrients; Dietary Supplement: Probiotic Yogurt A: Kaiser micronutrients; Dietary Supplement: Probiotic yogurt C: with basic micronutrients
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Probiotic Yogurt D: Placebo -- no added micronutrients

INTERVENTIONS:
Dietary Supplement: Probiotic Yogurt B: with various micronutrients — 175g probiotic yogurt / day 25% RDA for each nutrient
  Arms: 1
Dietary Supplement: Probiotic Yogurt A: Kaiser micronutrients — 175g probiotic yogurt/ day 25% RDA for each nutrient
  Arms: 1
Dietary Supplement: Probiotic yogurt C: with basic micronutrients — 175g yogurt/ day 25% RDA for each nutrient
  Arms: 1
Dietary Supplement: Probiotic Yogurt D: Placebo -- no added micronutrients — 175g/day probiotic yogurt
  Arms: 2

SUMMARY:
We hypothesize that micronutrient fortified probiotic yogurt can improve nutritional status and enhance immunity parameters in subjects HIV/AIDS and other immunodeficiencies.

We have developed a micronutrient-fortified probiotic yogurt that has safe and beneficial levels of micronutrients for human consumption. This has been undertaken with the guidance of Edward Farnworth, a senior research scientist at Agri-Food Canada-Food Research and Development Centre, St. Hyacinthe, Quebec

We will now measure nutritional parameters (height, weight, serum albumin, serum nutrient levels, blood urea, liver function tests (AST, ALT)) to determine if there is a statistically significant difference between the various levels of fortified probiotic yogurt and the placebo on the nutritional parameters of the subjects consuming the yogurt.

We will measure immunological parameters (CD4 lymphocyte count, CBC, levels of TNFα, IL-12, IL-10, and G-CSF [Kim, et.al. 2006]) in order to determine if there is a statistically significant difference using fortified probiotic yogurt compared to a placebo.

In addition, we will determine if the micronutrient-fortified probiotic yogurt has a significant impact on the overall quality of life for the subjects using the "linear analogue self assessment" tool [Kaiser, et.al 2006].

DETAILED DESCRIPTION:
Drs. Reid and Hekmat have recently developed a fermented milk product (yogurt) containing Lactobacillus GR-1 and RC-14 and concluded that such dairy products are suitable vehicles for these beneficial microorganisms [Hekmat, S. & Reid, G. 2006].

The strains Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 have a proven efficacy to treat and protect against gastrointestinal and urogenital infections [Anukam, K. et. al. 2006; 2007]. In one study, the supplementation of yogurt with these probiotics was shown to eradicate diahrea and increase the CD4 T-lymphocyte counts in HIV subjects [Anukam, K. et.al. 2006]. HIV infected subjects often suffer diarrheal episodes, and consequently experience malabsorption of certain nutrients [Cunningham-Rundles, 2000]. A study conducted by Cunningham et. al [2000] found that probiotic Lactobacillus plantarum 299 had a positive impact on the immunity of 10/17 children and on the growth of all of the children who were HIV-positive.

It is estimated that 75 percent of immune function is localized in the gastrointestinal tract, which may explain why oral administration of probiotics is an excellent tool for immunomodulation [Olah, A. et. al. 2002]. In a study of 45 patients with acute pancreatitis, 22 were given probiotic Lactobacillus plantarum 299 and 10g of oat fibre with regular enteral nutrition; and 23 were given a placebo in the form of regular enteral nutrition. Significantly fewer (n=1 versus n=7) patients in the probiotic/fibre group experienced septic complications requiring surgery, highlighting the safety and potential hospitalized benefits that could be accrued for critical care nutrition.

A study has recently shown in 40 HIV-infected patients taking a stavudine and/or didanosine-based HAART regimen plus micronutrients twice daily for twelve weeks, that the absolute CD4 count increased by an average of 24% versus 0% in the placebo group (p=0.01). The mean HIV-1 RNA decreased in the micronutrient supplementation group [Kaiser, et.al. 2006]. This is significant for the HIV/AIDS pandemic in Africa and for the many people in Canada living with HIV/AIDS. In addition, this may be related to other immunodeficiencies in hospitalized patients from chemotherapeutic and radiological treatments, organ transplantation, controlling diabetes, and other chronic ailments.

Clinical malnutrition is a heterogenous group of disorders including macronutrient deficiencies that lead to body cell mass depletion and micronutrient deficiencies, and these often coexist with infectious and inflammatory processes [Hughes,S. & Kelly, P. 2006]. Diverse factors affect bioavailability, such as the nutritional status of individuals, the presence in the diet of substances which facilitate or inhibit its absorption, interactions among micronutrients, illnesses, and chemical characteristics of the compound used for fortification. There is good evidence that specific micronutrients, particularly zinc and vitamin A, influence immunity, while iron supplementation is often not effective in Africa [Hughes, S. & Kelly, P. 2006].

More than 20% of older adults may have marginal or frank vitamin B12 deficiency [Park, et.al. 2006], while folic acid is often deficient in children and reproductive aged females. Glutamine, arginine, fatty acids, and vitamin E provide additional benefits to immunocompromised persons or patients who suffer from various infections, while long-chain polyunsaturated n-3 fatty acids, vitamin E, vitamin C, selenium, and nucleotides can modulate immunity to fight infection [Field, et.al. 2002]. In order to produce energy, the use of glucose by nervous tissue requires vitamin B1; this vitamin modulates cognitive performance, especially in the elderly. Vitamin B9 preserves brain during its development and memory during ageing. Vitamin B6 is likely to benefit in treating premenstrual depression. Vitamins B6 and B12, among others, are directly involved in the synthesis of some neurotransmitters [Bourre, JM. 2006]. Thus, three formulations added to L. rhamnosus GR-2 supplemented yogurt, will be tested at the Brescia College Tasting Centre where volunteers will score the products for taste and texture [Hekmat, S. & Reid, G. 2006]

Thirty test subjects will be recruited during the first four months of the study, for inclusion in a trial starting at the 4-6 month time-point, with completion by 10-12 months. A crossover study will be performed in London in which 10 HIV positive volunteers with CD4 counts between 200 and 400 on their standard treatment (including Highly Active Antiretroviral Therapy), and 10 subjects with Cancer who are in the recovery stages and not currently receiving chemotherapy or radiation therapy, and 10 healthy adults (aged 18-30) will randomly be assigned to receive one cup of Yogurts 1, 2 or 3 and a control unsupplemented yogurt 4, daily for one month, followed by a two week washout where no yogurt will be consumed, then one month on the second yogurt, two weeks off etc for 162 days. Subjects will not be receiving antibiotics, not have any mental illness that would affect compliance, or not be requiring surgery during the study. No restrictions will be placed on subjects continuing prescribed or other remedies, but none will consume any other probiotic product during the study. The volunteers will be gender matched and a randomization scheme will ensure that subjects are blinded and different yogurts are distributed at each time (thus, for example two subjects will receive yogurt 1, two yogurt 2, three yogurt 3 and three yogurt 4 on day sample day one). The two week washout period will be used, as probiotic organisms do not persist for longer than that. Various measurements will be taken on the day of consuming the first and last batches of yogurt (days 0, 30, 44, 74, 88, 118, 132, 162). These will include weight, height, and from blood samples the CD4 count, CBC, levels of TNFα, IL-12, IL-10 and G-CSF [Kim, et.al. 2006], liver function test (AST, ALT), serum albumin, total protein, blood urea, serum zinc levels, serum selenium levels and HIV-1 RNA. A linear analogue self-assessment tool will be used to assess the subject's energy levels, daily activities and overall quality of life [Kaiser, et.al. 2006].

The present project is an important step in developing new yogurts, supplemented with micronutrients and probiotic lactobacilli for malnourished children, adults, and seniors in Canada, as well as surgical, transplant, and hospitalized patients, and HIV/AIDS subjects in Canada and in Africa. The following formulations will be used to supplement the yogurt:

1. The Kaiser micronutrient formula [14]: N-Acetyl cysteine (NAC) 300 mg, Acetyl L-carnitine 250 mg, Magnesium 92.5 mg, Alpha lipoic Acid 100 mg, Selenium 13.8 µg, Beta carotene + Vitamin A 5666 IU, Zinc 2.4 mg, Vitamin C 21 mg, Copper 0.225 mg, Vitamin B1 0.3 mg, Boron 0.5 mg, Vitamin B2 0.3 mg, Potassium 1200 mg, Pantothenic acid 1.3 mg, Iron 3.3 mg, Niacinamide 3.8 mg, Manganese 0.5 mg, Inositol 15 mg, Biotin 7.5 µg, Vitamin B6 0.3 mg, Chromium 7.5 µg, Vitamin B12 0.6 µg, Molybdenum 11.3 µg, Vitamin D 52 IU, Choline 121.9 mg, Vitamin E 5.7 IU, Bioflavonoid complex 75 mg, Folic acid 100 µg, L-Glutamine 25 mg, Betaine HCL 37.5 mg;
2. A multi-component formula containing zinc 30mg, vitamins A + beta carotene 5666 IU , C 21mg and E 5.7 IU, selenium 13.8µg, iron 3.3mg, folic acid 100µg, vitamin B12 0.6 µg, vitamin B6 0.3 mg, vitamin B1 0.3mg
3. A basic supplement containing zinc 30mg, vitamins A 666 IU, vitamin C 21mg and E 5.7 IU, and folic acid 100µg and 16 mg docosahexaenoic acid (DHA-Omega 3 Fatty Acid) and 24mg eicosapentaenoic acid (EPA-Omega 3 Fatty Acid) [Austin, J. et.al 2006 & Alan DD, et.al 2006].

ELIGIBILITY:
Inclusion Criteria:

* Clinically tested CD4 lymphocyte count between 200-400cells/mL (HIV population)
* Confirmed cancer by physician (cancer population)
* Confirmed HIV by physician (HIV population)

Exclusion Criteria:

* Opportunistic infection
* Mental illness impairing ability to comply with study
* Pregnancy
* Currently consuming micronutrient supplement or probiotic
* Clinical history of lactose-intolerance or cow's milk allergies
* Require surgery, radiation or chemotherapy during the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09-07 (Actual); Primary Completion 2009-03-02 (Actual); Study Completion 2009-03-02 (Actual)

PRIMARY OUTCOMES:
Statistically significant improvement of immune status (CD4) Statistically significant improvement of nutritional status | Baseline and Follow-up for each yogurt type

SECONDARY OUTCOMES:
Improved quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Reid, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Dangour AD, Clemens F, Elbourne D, Fasey N, Fletcher AE, Hardy P, Holder GE, Huppert FA, Knight R, Letley L, Richards M, Truesdale A, Vickers M, Uauy R. A randomised controlled trial investigating the effect of n-3 long-chain polyunsaturated fatty acid supplementation on cognitive and retinal function in cognitively healthy older people: the Older People And n-3 Long-chain polyunsaturated fatty acids (OPAL) study protocol [ISRCTN72331636]. Nutr J. 2006 Aug 31;5:20. doi: 10.1186/1475-2891-5-20. PMID 16945130
- [Background] Anukam K, Osazuwa E, Ahonkhai I, Ngwu M, Osemene G, Bruce AW, Reid G. Augmentation of antimicrobial metronidazole therapy of bacterial vaginosis with oral probiotic Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14: randomized, double-blind, placebo controlled trial. Microbes Infect. 2006 May;8(6):1450-4. doi: 10.1016/j.micinf.2006.01.003. Epub 2006 Mar 29. PMID 16697231
- [Background] Anukam KC, Osazuwa EO, Osadolor HB, Bruce AW, Reid G. Yogurt containing probiotic Lactobacillus rhamnosus GR-1 and L. reuteri RC-14 helps resolve moderate diarrhea and increases CD4 count in HIV/AIDS patients. J Clin Gastroenterol. 2008 Mar;42(3):239-43. doi: 10.1097/MCG.0b013e31802c7465. PMID 18223503
- [Background] Austin J, Singhal N, Voigt R, Smaill F, Gill MJ, Walmsley S, Salit I, Gilmour J, Schlech WF 3rd, Choudhri S, Rachlis A, Cohen J, Trottier S, Toma E, Phillips P, Ford PM, Woods R, Singer J, Zarowny DP, Cameron DW; CTN 091/CRIT Cartenoids Study Group. A community randomized controlled clinical trial of mixed carotenoids and micronutrient supplementation of patients with acquired immunodeficiency syndrome. Eur J Clin Nutr. 2006 Nov;60(11):1266-76. doi: 10.1038/sj.ejcn.1602447. Epub 2006 May 24. PMID 16721396
- [Background] Bourre JM. Effects of nutrients (in food) on the structure and function of the nervous system: update on dietary requirements for brain. Part 1: micronutrients. J Nutr Health Aging. 2006 Sep-Oct;10(5):377-85. PMID 17066209
- [Background] Cunningham-Rundles S, Ahrne S, Bengmark S, Johann-Liang R, Marshall F, Metakis L, Califano C, Dunn AM, Grassey C, Hinds G, Cervia J. Probiotics and immune response. Am J Gastroenterol. 2000 Jan;95(1 Suppl):S22-5. doi: 10.1016/s0002-9270(99)00813-8. PMID 10634225
- [Background] Field CJ, Johnson IR, Schley PD. Nutrients and their role in host resistance to infection. J Leukoc Biol. 2002 Jan;71(1):16-32. PMID 11781377
- [Background] Hekmat, S & Reid, G. 2006 The survival of Lactobacillus reuteri RC-14 and Lactobacillus rhamnosus GR-1 in milk. International Journal of Food Science and Technology (in press).
- [Background] Hughes S, Kelly P. Interactions of malnutrition and immune impairment, with specific reference to immunity against parasites. Parasite Immunol. 2006 Nov;28(11):577-88. doi: 10.1111/j.1365-3024.2006.00897.x. PMID 17042929
- [Background] Kaiser JD, Campa AM, Ondercin JP, Leoung GS, Pless RF, Baum MK. Micronutrient supplementation increases CD4 count in HIV-infected individuals on highly active antiretroviral therapy: a prospective, double-blinded, placebo-controlled trial. J Acquir Immune Defic Syndr. 2006 Aug 15;42(5):523-8. doi: 10.1097/01.qai.0000230529.25083.42. PMID 16868496
- [Background] Kim SO, Sheikh HI, Ha SD, Martins A, Reid G. G-CSF-mediated inhibition of JNK is a key mechanism for Lactobacillus rhamnosus-induced suppression of TNF production in macrophages. Cell Microbiol. 2006 Dec;8(12):1958-71. doi: 10.1111/j.1462-5822.2006.00763.x. Epub 2006 Aug 2. PMID 16889627
- [Background] Olah A, Belagyi T, Issekutz A, Gamal ME, Bengmark S. Randomized clinical trial of specific lactobacillus and fibre supplement to early enteral nutrition in patients with acute pancreatitis. Br J Surg. 2002 Sep;89(9):1103-7. doi: 10.1046/j.1365-2168.2002.02189.x. PMID 12190674
- [Background] Park S, Johnson MA. What is an adequate dose of oral vitamin B12 in older people with poor vitamin B12 status? Nutr Rev. 2006 Aug;64(8):373-8. doi: 10.1111/j.1753-4887.2006.tb00222.x. PMID 16958314
- See also: Canadian Research and Development Centre for Probiotics — http://www.crdc-probiotics.ca/